CLINICAL TRIAL: NCT05078502
Title: Role of Vitamin D3 Supplementation With Conventional Synthetic Disease Modifying Antirheumatic Drugs (csDMARD) in Rheumatoid Arthritis Patients: Randomized Double-blind Placebo Controlled Trial
Brief Title: Role of Vitamin D3 Supplementation With Conventional Synthetic Disease Modifying Antirheumatic Drugs(csDMARD) in Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Sultana Aktia Islam, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2021/3958
Record Dates: First submitted 2021-10-04; First posted 2021-10-14 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Immediately after randomization, random numbers of the two sets were assigned as patient code number. One set was designated as intervention group and another set was placebo group. Then the set of code numbers that belong to the intervention group were written as patient ID numbers on the packages contained vitamin D3 capsules. On the other hand, the set belongs to the placebo group were designated as patient ID numbers on the packages containing placebo capsules. This total procedure was conducted by the persons unrelated to this research. Thus the participants, caregiver, outcome assessor and the analyst, who require being blind for such study, were effectively blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Vitamin D3 along with CsDMARDs (Active Comparator): One capsule of vitamin D3 (40000IU) weekly for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3
- Placebo of Vitamin D3 along with CsDMARDs (Placebo Comparator): One capsule of placebo of vitamin D3(40000IU) weekly for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — One capsule of vitamin D3(40000IU) weekly for 8 weeks

SUMMARY:
Several studies suggested low serum level of vitamin D have been associated with rheumatoid arthritis. So, the present study was designed to investigate the effect of vitamin D supplementation along with CsDMARD in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory autoimmune disease that causes synovitis in the peripheral joints as well as extra-articular symptoms. With a good response to conventional drugs, treatment for this disease remains unsatisfactory. Vitamin D deficiency is now widely recognized as a problem in RA patients. Some recent trials have attempted to analyze the effect of vitamin D3 supplementation on pain intensity and disease activity in patients, and the majority of them have found significant improvement. The goal of this trial was to see if supplementing vitamin D3 with conventional synthetic DMARDs improved the intensity of pain and disease activity in RA patients. This study was a randomized, double-blind, placebo-controlled trial and was conducted in the Department of Pharmacology, BSMMU in collaboration with the Rheumatology Rehabilitation Clinic of the Department of Physical Medicine and Rehabilitation, BSMMU. Patients were assessed using a validated version of the visual analog scale (VAS) and the DAS-28 CRP scale. A total of 58 RA patients were selected based on inclusion and exclusion criteria, and baseline CRP levels were measured serum preserved for vitamin D3 estimation. A physiatrist at the Physical Medicine and Rehabilitation department's Rheumatology Rehabilitation Clinic performed the clinical diagnosis of RA patients. Following the completion of the necessary formalities, including the patients' informed consent, the patient has given a Visual Analog Scale (VAS) questionnaire to assess pain improvement and a disease activity score -28 C-Reactive Protein (DAS-28 CRP) scale to assess disease activity. The patients were split into two arms at random: intervention and control. Patients in the intervention arm received csDMARDs plus vitamin D3 (40,000IU) for 8 weeks. Weekly oral vitamin D3 (40,000IU) was given to the intervention arm. On the other hand, The placebo arm got csDMARD in the form of one oral placebo capsule once a week for the same duration of time. After 8 weeks of therapeutic intervention, blood samples were taken to determine serum 25 hydroxyvitamin D and CRP levels. The baseline and after 8 weeks serum 25 hydroxyvitamin D levels were estimated at the same time. The patient's compliance sheet, as well as the phone and pill count, were used to verify that medicine intake was regular. Microsoft Office Excel 2007 was used to perform the statistical analysis. A chi-squared test was used to analyze the relationship between the intervention and placebo arms. An unpaired t-test was used to compare the scores of the two arms. A paired t-test was employed to compare the score before and after the intervention. A total of 58 people were enrolled in this study over six months. Following decoding, it was established that twenty-nine (30) patients would receive vitamin D3 and twenty-three (28) would receive a placebo. Among them, fifty-two (52) patients met all criteria to be eligible for analysis. There was a substantial difference in improving disease activity and pain severity between the two arms (p-value- 0.00). All of the RA patients were vitamin D deficient. Vitamin D3 supplementation for 8 weeks resulted in a significantly higher level than the placebo arm (p- 0.01), as well as a significant increase from the baseline level (p- 0.04). After 8 weeks of vitamin D3 administration, CRP levels were significantly reduced (p-0.00). There was no correlation between serum 25-hydroxyvitamin D levels and disease activity. Vitamin D3 significantly reduced the intensity of pain and disease activity in conventional synthetic Disease-Modifying Antirheumatic Drugs (csDMARD) treated Rheumatoid Arthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met 2010 ACR/EULAR criteria for Rheumatoid arthritis
* Age: 18 years or above
* Both gender

Exclusion Criteria:

* Overlapped syndrome
* Patients with renal and liver disease, malabsorption, hyperparathyroidism
* Spondyloarthritis, psoriatic arthritis, Systemic lupus erythematosus
* Patients receiving vitamin D3, anti TB like rifampicin, isoniazid, anti-seizure drugs within last two months
* Patients unwilling to participate or unwilling to give written consent
* Pregnant & lactating woman
* Impaired cognitive function

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Severity of pain | 8 weeks
  Changes in severity of pain will be measured through the Visual Analog Scale (VAS) at baseline and at 8 weeks, minimum value 0 and maximum value 10, higher score mean a worse outcome.
Disease activity | 8 weeks
  Changes in DAS-28-CRP score between placebo and intervention arm at baseline and after 8 weeks of treatment by DAS-28-CRP scale

SECONDARY OUTCOMES:
measure serum 25 hydroxyvitamin D level | 8 weeks
  To compare the serum 25- Hydroxyvitamin D level between placebo and intervention arm at baseline and after 8 weeks of treatment
C- Reactive Protein Level | 8 weeks
  To compare the serum C-reactive protein level between placebo and intervention arm at baseline and after 8 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Md. Sayedur Rahman, MBBS, Mphil, FCPS, Study Chair — BSMMU, Bangladesh
Locations (1):
- BSMMU, Dhaka, Bangladesh